CLINICAL TRIAL: NCT02619578
Title: The Effect of Transcutaneous Electric Acupoint Stimulation on the Quality of Early Recovery in Patients Undergoing Gynecological Laparoscopic Surgery: a Prospective, Randomized, Placebo-controlled Trial
Brief Title: The Effect of TEAS on the Quality of Early Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A14-30323
Record Dates: First submitted 2015-11-20; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: C.Delivery; Surgery (Previous), Gynecological; Inappropriate Device Stimulation of Tissue; Delayed Emergence From Anesthesia
Keywords: Transcutaneous electric acupoint stimulation (TEAS); gynecological laparoscopic surgery; QoQ-40; MMSE; VAS
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Propofol; Remifentanil; Vecuronium Bromide; Respiration, Artificial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEAS Group (Other): TEAS consisted of 30 min of stimulation (12-15 mA, 2/100 Hz) at the Hegu (L14) and Neiguan (PC6) before anesthesia. Anesthesia was induced i.v. with propofol (2 mg kg-1) and remifentanil (1 μg kg-1) using a target-controlled infusion (TCI) system. After loss of consciousness, vecuronium (0.1 mg kg-1) was administered i.v. Patients' lungs were mechanically ventilated in a volume-controlled mode with a tidal volume of 8ml kg-1 body weight during the operation.
  Interventions: Other: TEAS; Drug: propofol, remifentanil, vecuronium; Other: mechanical ventilation
- Con Group (Other): The patients in the Con group had the electrodes applied at the same acupoints, but received no stimulation. Anesthesia was induced i.v. with propofol (2 mg kg-1) and remifentanil (1 μg kg-1) using a target-controlled infusion (TCI) system. After loss of consciousness, vecuronium (0.1 mg kg-1) was administered i.v. Patients' lungs were mechanically ventilated in a volume-controlled mode with a tidal volume of 8ml kg-1 body weight during the operation.
  Interventions: Other: Con; Drug: propofol, remifentanil, vecuronium; Other: mechanical ventilation

INTERVENTIONS:
Other: TEAS — According to the theory of traditional Chinese medicine, bilateral Baihui (GV20), Yingtang (EX-HN3), Zusanli (ST36) and Neiguan (PC6) were chosen as the acupuncture points. These acupoints were identified according to the traditional anatomic localization . Gel electrodes were applied to the skin after it had been cleaned with ethyl alcohol. The acupoints were then stimulated electrically with an intensity of 12-15 mA and dense-disperse frequency of 2/100 Hz for 30 min, using the Hwato electronic acupuncture treatment instrument (model No. SDZ-V, Suzhou Medical Appliances Co., Ltd, Suzhou, China). The intensity was adjusted to maintain a slight twitching of local muscles according to individual maximum tolerance, indicating a satisfactory of De-Qi phenomenon and thus adequate stimulation.
  Arms: TEAS Group
Other: Con — The patients in the Con group had the electrodes applied at the same acupoints, but received no stimulation.
  Arms: Con Group
Drug: propofol, remifentanil, vecuronium — Anesthesia was induced i.v. with propofol (2 mg kg-1) and remifentanil (1 μg kg-1) using a target-controlled infusion (TCI) system. After loss of consciousness, vecuronium (0.1 mg kg-1) was administered i.v.
Other: mechanical ventilation — Patients' lungs were mechanically ventilated in a volume-controlled mode with a tidal volume of 8ml kg-1 body weight during the operation.

SUMMARY:
During the past four decades, gynecologic laparoscopy has evolved from a limited method to an advanced operative approach that frequently serves as a substitute for laparotomy. The advantages of laparoscopy over laparotomy include less postoperative pain, shorter hospital stays, and reduced blood loss. However, in the surgery CO2 increases the intra-abdominal and intrathoracic pressure, which leads to cardiac output decrease and increases sympathetic activity in a reflex. On the other hand, CO2 accumulation in the body leads to hypercapnia, which indirectly stimulates aortic body chemosensory organs and carotid sinus, increasing the concentration of plasma catecholamines, cortisol and vasopressin , these responses have an important impact on patient recovery after surgery.

Acupuncture is an ancient Chinese method to treat diseases and relieve pain. Transcutaneous electrical acupoint stimulation (TEAS), a noninvasive adjunctive intervention based on acupuncture, has been widely accepted and used worldwide. To date, multiple studies have demonstrated TEAS could reduce intra-operative opioid drugs consumption, reduce the incidence of postoperative nausea and vomiting (PONV) and improve postoperative cognitive function. However, whether TEAS could improve the quality of early recovery after gynecologic laparoscopy is unknown. In this study we therefore investigated the effects of TEAS at the acupoints of Baihui (GV20), Yingtang (EX-HN3), Zusanli (ST36) and Neiguan (PC6) on the quality of early recovery in the patients undergoing gynecological laparoscopic surgery.

DETAILED DESCRIPTION:
Patient population Sixty patients undergoing elective gynecological laparoscopic surgery at Guizhou province people's hospital with an ASA physical status of I-II were recruited between November 2013 and November 2014. Their ages ranged from 29-60 yr. Exclusion criteria were recent use of TEAS or acupuncture, neural damage or infection along the meridian at which the acupoints lay, use of antiemetic in the previous week, regular use of opioids, hepatic dysfunction, confirmed renal impairment, diabetes mellitus, cognitive dysfunction and conversion to laparotomy during gynecologic laparoscopy.

Randomization and blinding Patients were assigned to either TEAS stimulus (TEAS group) or control group (Con group) on the basis of random numbers generated by a computer. Only the acupuncturist was informed the randomization allocation, just before the onset of TEAS. None of the anesthesiologists, surgeons, physicians in the post-anesthesia care unit (PACU), or participants were aware of the allocation. Blinding of the patients was ensured by using gel electrodes in the same therapeutic setting, which has previously been proved to be a successful strategy.

TEAS protocol An experienced acupuncturist performed TEAS for 30 min before anesthesia. According to the theory of traditional Chinese medicine, bilateral Baihui (GV20), Yingtang (EX-HN3), Zusanli (ST36) and Neiguan (PC6) were chosen as the acupuncture points. These acupoints were identified according to the traditional anatomic localization. Gel electrodes were applied to the skin after it had been cleaned with ethyl alcohol. The acupoints were then stimulated electrically with an intensity of 12-15 mA and dense-disperse frequency of 2/100 Hz for 30 min, using the Hwato electronic acupuncture treatment instrument (model No. SDZ-V, Suzhou Medical Appliances Co., Ltd, Suzhou, China). The intensity was adjusted to maintain a slight twitching of local muscles according to individual maximum tolerance, indicating a satisfactory of De-Qi phenomenon and thus adequate stimulation. The patients in the control group had the electrodes applied but received no stimulation.

Anesthesia and perioperative management One surgeon conducted all surgeries according to a standard protocol; surgery commenced between 8:30 and 1:00 p.m. Anesthesia was induced i.v. with propofol and remifentanil using a target-controlled infusion (TCI) system. After loss of consciousness, vecuronium (0.1 mg kg-1) was administered i.v., and patients were orotracheally intubed 5 min later. Anesthesia was maintained with TCI of propofol and remifentanil. The depth of anesthesia was monitored using index (BIS). Effect site concentrations of propofol and remifentanil were adjusted to the hemodynamic and BIS. Patients' lungs were mechanically ventilated in a volume-controlled mode with a tidal volume of 8ml kg-1 body weight during the operation. In both groups, remifentanil and propofol infusions were stopped 5 min before the end of surgery. Patients were extubated and transferred to the PACU after surgery.

Data collection Baseline data included demographics, body mass index (BMI), and ASA physical status. Surgical information recorded included anesthesia duration, surgery duration, estimated blood loss, and all other intraoperative medications. Postoperative data were collected regarding the incidence of nausea and vomiting, postoperative pain medications and antiemetics.

The Quality of Recovery-40 (QoR-40) is a validated scale with 5 domains 10-12. These measure physical comfort, emotional state, physical independence, psychological support, and pain. Each domain is scored to a maximum global score of 200. QoR-40 scores have been found to be associated with both quality-of-life scales and patient satisfaction indices 13 as well as postoperative pain 14. In the present study, QoR-40 evaluation was performed on preoperative day 1(T0), postoperative day 1 (T1) and postoperative day 2 (T2).

Visual analog scales (VAS) are widely used in behavioral science and previous studies reported their usefulness and validity 15, 16. VAS scores at rest queried about their level of pain on postoperative day 1 (T1) and postoperative day 2 (T2).

The Mini-Mental State Examination (MMSE) is one of the most widely used assessment instruments of cognitive functioning postoperatively, which screens domains of orientation to time and place, attention and memory, concentration, language and praxis 17. Patient cognitive function was assessed using the MMSE on preoperative day 1(T0), postoperative day 1 (T1) and postoperative day 2 (T2).

Statistical analysis All statistical analyses were performed using SPSS 13.0 (SPSS, Inc., Chicago, IL, USA). Continuous variables are presented as mean (SD) and compared using the unpaired Student's-test. Dichotomus variables were presented as the number of patients (percent) and analyzed using the X2 test. The level of significance for all statistical tests was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective gynecological laparoscopic surgery.
* ASA physical status of I-II.
* Ages ranged from 29-60 yr.

Exclusion Criteria:

* Recent use of TEAS or acupuncture.
* Neural damage or infection along the meridian at which the acupoints lay.
* Use of antiemetic in the previous week.
* Regular use of opioids.
* Hepatic dysfunction.
* Confirmed renal impairment. Diabetes mellitus Cognitive dysfunction Conversion to laparotomy during gynecologic laparoscopy.

Ages: 29 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Scores on QoR-40 | 1 year
  Quality of recovery was assessed using a 40-item questionnaire as a measure of quality of recovery (QoR-40; maximum score 200) scoring system performed on preoperative day 1(T0), postoperative day 1 (T1) and postoperative day 2 (T2).

SECONDARY OUTCOMES:
Scores on MMSE | 1 year
  mini-mental state examination (MMSE) scores performed on preoperative day 1(T0), postoperative day 1 (T1) and postoperative day 2 (T2).
Scores on VAS | 1 year
  A 100-mm visual analogue scale (VAS) scores at rest performed on preoperative day 1(T0), postoperative day 1 (T1) and postoperative day 2 (T2).

OTHER OUTCOMES:
The incidence of nausea and vomiting | 1 year
  The incidence of nausea and vomiting were also recorded.Nausea was defined as a subjective unpleasant sensation associated with awareness of the urge to vomit; vomiting was defined as the forceful expulsion of gastric contents from the mouth brought about by the powerful sustained contraction of abdominal muscles.
The incidence postoperative pain medications | 1 year
  The incidence of postoperative pain medications were recorded.
The incidence postoperative antiemetics | 1 year
  The incidence of antiemetics were also recorded.
Age | 1 year
  The patients' age were recorded
Height | 1 year
  The patients' height were recorded
Body mass index (BMI) | 1 year
  The patients' BMI were recorded
ASA physical status | 1 year
  ASA physical status of patients were recorded
Anesthesia duration and surgery duration | 1 year
  Anesthesia duration was recorded
Intra-operative fluids | 1 year
  Intra-operative fluids was recorded

REFERENCES:
- [Derived] Yu X, Zhang F, Chen B. The effect of TEAS on the quality of early recovery in patients undergoing gynecological laparoscopic surgery: a prospective, randomized, placebo-controlled trial. Trials. 2020 Jan 8;21(1):43. doi: 10.1186/s13063-019-3892-4. PMID 31915045